CLINICAL TRIAL: NCT01462851
Title: A Phase 1, Randomized Investigator-And-Subject-Blind, Sponsor Open, Placebo Controlled Two-Part Study To Characterize The Pharmacokinetics And Pharmacodynamics Of Single Doses Of Pf-05297909 In Healthy Adult Subjects
Brief Title: A Study To Observe Safety And Concentrations Of PF-05297909 And Proteins In Both Blood And Cerebrospinal Fluid After A Single Dose Of PF-05297909 In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B3941001
Record Dates: First submitted 2011-09-08; First posted 2011-10-31 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: healthy volunteer; safety; pharmacokinetic; pharmacodynamic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation (Experimental): Ascending doses in healthy volunteers
  Interventions: Drug: PF-05297909 25 mg; Drug: PF-05297909 100 mg; Drug: PF-05297909 250 mg; Drug: PF-05297909 525 mg
- Part 2: CSF PKPD (Experimental): Pharmacokinetic and pharmacodynamic cerebrospinal fluid assessment
  Interventions: Drug: PF-05297909 525 mg

INTERVENTIONS:
Drug: PF-05297909 25 mg — Single oral (PO) dose, PF-05297909 25 mg
  Arms: Dose Escalation
Drug: PF-05297909 100 mg — Single oral (PO) dose, PF-05297909 100 mg
  Arms: Dose Escalation
Drug: PF-05297909 250 mg — Single oral (PO) dose, PF-05297909 250 mg
  Arms: Dose Escalation
Drug: PF-05297909 525 mg — Single oral (PO) dose, PF-05297909 525 mg
  Arms: Dose Escalation
Drug: PF-05297909 525 mg — Single oral (PO) dose, 525 mg
  Arms: Part 2: CSF PKPD

SUMMARY:
This study is designed to observe the safety and concentrations of PF-05297909 and proteins in both blood and cerebrospinal fluid after a single dose of PF-05297909 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* For Healthy adult volunteers: healthy male and/or female subjects of non child bearing potential between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests.)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Plasma area under the curve last (AUClast) pharmacokinetic parameter | Day 1 to Day 3
Plasma apparent clearance (CL/F) pharmacokinetic parameter | Day 0 to Day 3
Clinical potency of PF 05297909 for reduction in CSF levels of Abeta40, Abeta42, and/or AbetaX via estimation of the IC50 from a population PK/PD (PPK/PD) model | Day 0 to Day 3
Plasma area under the curve infinity (AUCinf) pharmacokinetic parameter | Day 1 to Day 3
Plasma half-life (t1/2) pharmacokinetic parameter | Day 1 to Day 3
Plasma apparent volume of distribution (Vz/F) pharmacokinetic parameter | Day 1 to Day 3
CSF concentration summary by time point for PF 05297909. | Day 1 to Day 3
Change from baseline in CSF levels of Abeta40 | Day 1 to Day 3
Change from baseline in CSF levels of Abeta42 | Day 1 to Day 3
Change from baseline in CSF levels of AbetaX | Day 1 to Day 3
Change from baseline in CSF levels of sAPPalpha | Day 1 to Day 3
Change from baseline in CSF levels of sAPPbeta. | Day 1 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, New Haven, Connecticut

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3941001&StudyName=A%20Study%20To%20Observe%20Safety%20And%20Concentrations%20Of%20PF-05297909%20And%20Proteins%20In%20Both%20Blood%20And%20Cerebrospinal%20Fluid%20After%20A%20Single%20Dose%20O